CLINICAL TRIAL: NCT02715154
Title: Effect and Placental Transfer of Dexmedetomidine During Caesarean Section Under Epidural Anaesthesia
Brief Title: Dexmedetomidine for Cesarean Section
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Cunming Liu, Chief officer, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: JSPH-A-1
Record Dates: First submitted 2016-03-02; First posted 2016-03-22 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Cesarean Section, Affecting Fetus or Newborn
Keywords: Epidural Anaesthesia; Cesarean Section; Dexmedetomidine
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine 0.5 µg/kg/h (Active Comparator): Solution containing 5 µg/mL of dexmedetomidine was continuously infused by 0.5 μg/kg in 10 min, followed with 0.1 ml/kg/hr continuous infusion until the closure of the abdominal.
  Interventions: Drug: Dexmedetomidine
- Placebo (Placebo Comparator): The placebo group (n = 20) will pumped in the same volume of saline 0.9% as calculated by patients' weight in 10 min, then will receive an i.v. infusion of 0.1 mL/kg/h saline 0.9%, until the closure of the abdominal.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexmedetomidine — The dexmedetomidine groups (n = 20 ) will receive i.v. infusion of 0.5 μg/kg of solution containing 5 µg/mL of dexmedetomidine, at 10 min after the level of anesthesia completed. Followed with 0.1ml/kg/hr continuous infusion until the closure of the abdominal.The placebo and the dexmedetomidine solutions will be looked identical and their infusions will be continued until skin closure.
  Other Names: Dexmedetomidine Hydrochloride Injection
  Arms: Dexmedetomidine 0.5 µg/kg/h
Drug: Placebo — The placebo group (n = 20) will pumped in the same volume of saline 0.9% as calculated by patients' weight in 10 min, then will receive an i.v. infusion of 0.1 mL/kg/h saline 0.9%, until the closure of the abdominal. The placebo and the dexmedetomidine solutions will be looked identical and their infusions will be continued until skin closure.
  Arms: Placebo

SUMMARY:
Current cesarean section often chooses spinal anesthesia. And in order to avoid the impact of drugs on the fetus, before the delivery, anesthesiologist generally don't use sedative or analgesic drugs. However, the majority of puerperas would appear nervous, anxiety, fear and other psychological reactions in cesarean section. Although the placental transfer and the foetal metabolism of dexmedetomidine have been reported and the result show no adverse effects on neonates, but the placental transfer of dexmedetomidine in intravertebral anesthesia area was lack of systematical research. This study intends to use of dexmedetomidine in the cesarean section under epidural anesthesia and investigate its effects on the parturients' haemodynamics and the neonates' placental transfer and metabolism.

DETAILED DESCRIPTION:
Current cesarean section in domestic and overseas often chooses spinal anesthesia. And in order to avoid the impact of drugs on the fetus, before the delivery, anesthesiologist generally don't use sedative or analgesic drugs. However, the majority of puerperas would appear nervous, anxiety, fear and other psychological reactions in cesarean section, and thus produced a series of stress reactions that not only cause the hemodynamic fluctuating in anesthesia and operation, but also lead to different degrees of personality and behavior changed. It causes serious injury to physical and mental health of patients. Dexmedetomidine is a highly selective α2 receptors agonist (α2-AR) ，it has sedation, analgesia, antisympathetic pharmacological effects and unique "conscious sedation" without respiratory depression. At present, dexmedetomidine has been widely used in patients in clinics and clinical anesthesia, it has been hailed as an"dvocate medicine in modern comfortable anesthesia."Experiments in animals have shown that dexmedetomidine had no adverse effects on pregnant rats. In addition, Dexmedetomidine has successful application in preterm infants, infants and children anesthesia, also has a few for caesarean patients sedation reports. Although the placental transfer and the foetal metabolism of dexmedetomidine have been reported and the result show no adverse effects on neonates, but the placental transfer of dexmedetomidine in intravertebral anesthesia area was lack of systematical research.

The safety of the use of dexmedetomidine on neonatal outcome is a very important issue. Experimental study on acute exposure of rats to dexmedetomidine at the anticipated delivery time recorded absence of any adverse effects on perinatal morphology of pups, their birth weight, crown-rump length, physical growth and postnatal behavioural performances. Others studied the transfer of clonidine and dexmedetomidine across the isolated perfused human placenta. Dexmedetomidine disappeared faster than clonidine from the maternal circulation, while even less dexmedetomidine was transported into the fetal circulation. This was due to its greater placental tissue retention, the basis for which probably is the higher lipophilicity of dexmedetomidine.

Umbilical cord blood gas analysis of umbilical vein and umbilical artery in this study was similar to the results of previous studies . The partial oxygen pressure (PO2) of the arterial blood gas in the umbilical vein was not significantly affected to the oxygen supply of the newborn infants. On the other hand, the umbilical arterial blood gas was the most reliable indicator of the oxygenation index and acid-base status of the fetus. Previous studies have indicated that the relationship between hydrogen ion concentration(PH), base excess（BE） and neonatal asphyxia was relatively large, and it was positively related to growth.

Previous research of in vitro placental perfusion indicated that the transfer rate of dexmedetomidine through the placenta to foetus was 0.77, and the other study indicated that the rate of placental transfer of dexmedetomidine in cesarean section operation under general anesthesia was 0.76. It's indicated that dexmedetomidine can also easily pass through the placental barrier like other anaesthetic drugs. However, the placental transfer rate of dexmedetomidine is much lower than that of clonidine(0.85) and that of remifentanil(0.88), which may be caused by dexmedetomidine being more fat-soluble and easier to be retained in the placenta.

Recently, there is a published interested case report about the successful use of dexmedetomidine 1 µg/kg followed with 1 µg/kg/h for 10 minutes before cesarean delivery to facilitate awake fiberoptic endotracheal intubation patient with spinal muscular atrophy type III with provided adequate sedation, without respiratory compromise. Although pharmacokinetic data cannot be determined, this case confirms existing in vitro data that dexmedetomidine has significant placental transfer. Nevertheless, serious neonatal effects were not detected. Similarly, others used, i.v. dexmedetomidine successfully as an adjunct to opioid-based PCA and general anesthesia for the respective provision of labor analgesia and cesarean delivery anesthesia in a parturient with a tethered spinal cord, with favourable maternal and neonatal outcome.

Project Objectives:

The investigators hypothesize that application of dexmedetomidine in cesarean section under epidural anesthesia was conducive to maintaining the stability of hemodynamics of the patients, reducing patients' anxiety and pain stress during the operations, which also had no adverse effects on newborns.

The aims of the present study are:

Our research efforts will focus on identifying the effects of 0.5 µg/kg/h dexmedetomidine for uncomplicated cesarean delivery on the followings.

Hemodynamic [heart rate, systolic and mean blood pressure] changes. The rate of placental transfer of dexmedetomidine . Apgar score (1 and 5 minute) after delivery. The umbilical cord venous and arterial blood gases analyses. The sedation of Dexmedetomidine. The incidence of the major complications (respiratory, cardiovascular events, nausea, vomiting and other adverse reactions).

Project Design:

Study Design:

The study was approved by the first affiliated hospital ethics committee of Nanjing Medical University, and the puerperas and their families signed informed consent.

Sampling Site:

I. Patient Selection: patients aged 23-41 years (ASA physical status I-II) scheduled for elective in about 40 women (American Society of Anesthesiologists [ASA] I and II), with uncomplicated, singleton pregnancies, who will receive epidural anesthesia. The investigators will exclude women with a history of cardiac, liver, or kidney diseases; allergy to amide local anesthetics; epilepsy; those taking cardiovascular medications; and those with pregnancy-induced hypertension, evidence of intrauterine growth restriction, or fetal compromise.

II. Anesthesia method

Routine monitoring such as electrocardiogram(ECG), heart rate(HR), saturation of pulse oxygen(SpO2) were monitored after patient arrived at the operation room. Selected the forearm vein to open venous access, infused sodium lactate Ringer's solution before anaesthesia. Then began to epidural anesthesia: The patients were at left side lying position, the L2,3 gap was chosen for puncture. After determined the success of puncture, inserted the epidural catheter into the head side, the length of the epidural space is 4cm. By intraductal injection of 2% lidocaine 3ml, signs of spinal anesthesia were excluded. Additional 0.75% ropivacaine 10 ~ 20ml was injected to control the level of pain disappear on thoracic4(T4) or thoracic6(T6) to satisfy the operation needs. After the level of anesthesia completed, Dex group: dexmedetomidine was continuously infused by 0.5 μg/kg in 10 min, followed with 0.5 μg/kg/hr continuous infusion until the closure of the abdominal. normal saline(NS)group: Pumped in the same volume of normal saline. In the operation, if the blood pressure was lower than 70% before anesthesia given ephedrine 10 ~ 15mg, and 0.5mg atropine was used when the heart rate was lower than 60 beats per minute. All operations were performed by the same group of maieutologists.

III. The Investigators who will be involved with subsequent postoperative patient assessment will be blinded of the patient group.

IV. Observational information

Systolic pressure(SBP) and diastolic blood pressure(DBP), heart rate(HR) were recorded at four time points: before anesthesia(T0), infused 10 min(T1), at the delivery of the baby(T2), at the end of the operation(T3). Ramsay sedation scales were evaluated at three time points: before anesthesia (T0), skin incision (T1) and 10min after delivery (T2). (Ramsay standard for evaluation: 1 point: anxious or restless or both; 2 point: cooperative, orientated and tranquil; 3 point: responding to commands; 4 point: brisk response to stimulus; 5 point: sluggish response to stimulus; 6 point: no response to stimulus. The Apgar scores were evaluated at 1 and 5 minute after the delivery. The urinary volume, the bleeding volume and the infusion volume during the operation were measured. Adverse effects such as nausea and vomiting in 24 hour after the operation were recorded. Postoperative analgesic formula: 12mg butorphanol tartrate, 9mg granisetron hydrochloride, diluted with normal saline to 100ml. Background dose: 2 milliliter per hour, patient controlled analgesia (PCA): 0.5 milliliter, locking time:15 minutes.

V. Samples Collection and Analysis For blood gas analysis and the plasma dexmedetomidine concentrations:

Maternal venous blood samples (MV), umbilical artery(UA) and umbilical vein(UV) will be collected for blood gas analysis, plasma dexmedetomidine concentrations. concentrations at points: When the baby was born.

1. Type of samples: centrifuged 3500 revolutions per minute for 5 minutes and separated of plasma to -20℃ frozen preservation.
2. Laboratory Analysis:

High-performance liquid chromatography-mass spectrometry(HPLC-MS/MS) was then used for measuring the plasma dexmedetomidine concentrations [concentration of umbilical vein(CUV), concentration of umbilical artery(CUA) and concentration of maternal vein(CMV)]..

VI. Statistical Analysis: The statistical analysis was performed with SPSS 22.0. The measurement data are shown as mean ± standard deviation (x±s), the t-test was used for comparison between the groups, and repeated measures analysis of variance was performed for comparison within the group; chi-square test was used for comparison of the count data, and rank-sum test was used for comparison of the level information. p < 0.05 was considered as statistically significant.

VII. Report Writing: 2 months

ELIGIBILITY:
Inclusion Criteria:

* 40 cases of full-term puerperas with single baby ASA I or II, aged 23 to 41 years old, weighing 61-92 kg, without spinal canal puncture contraindication and scheduled for caesarean section under epidural anesthesia were selected for this study.

Exclusion Criteria:

* women with a history of cardiac, liver, or kidney diseases;
* women with allergy to amide local anesthetics;
* women with epilepsy;
* those taking cardiovascular medications;
* those with pregnancy-induced hypertension;
* women with evidence of intrauterine growth restriction or fetal compromise.

Ages: 23 Years to 41 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-06; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Systolic blood pressure of Dexmedetomidine in Epidural Anaesthesia | before anesthesia, infused 10 min, at the delivery of the baby, at the end of the operation
  identifying the effects of 0.5 µg/kg/h dexmedetomidine for systolic blood pressure changes.
Diastolic blood pressure of Dexmedetomidine in Epidural Anaesthesia | before anesthesia, infused 10 min, at the delivery of the baby, at the end of the operation
  identifying the effects of 0.5 µg/kg/h dexmedetomidine for diastolic blood pressure changes.
Saturation of pulse oxygen of Dexmedetomidine in Epidural Anaesthesia | before anesthesia, infused 10 min, at the delivery of the baby, at the end of the operation
  identifying the effects of 0.5 µg/kg/h dexmedetomidine for saturation of pulse oxygen changes.
Heart rate of Dexmedetomidine in Epidural Anaesthesia | before anesthesia, infused 10 min, at the delivery of the baby, at the end of the operation
  identifying the effects of 0.5 µg/kg/h dexmedetomidine for heart rate changes.

SECONDARY OUTCOMES:
Apgar score related to treatment | 1 and 5 minute after delivery
  Apgar score：The Apgar scores were evaluated at 1 and 5 minute after the delivery.
Blood gas analysis | at the delivery of the baby
  The difference of blood gas analysis from MV, UA , UV.
adverse events | intraoperative and in 48 hours after surgery
  Major complications (respiratory, cardiovascular events, nausea, vomiting and other adverse reactions)
plasma concentrations of dexmedetomidine | at the delivery of the baby
  identifying the effects of 0.5 µg/kg/h dexmedetomidine for the plasma dexmedetomidine concentrations (CUV, CUA and CMV).
sedation of Dexmedetomidine in Epidural | before anesthesia, skin incision and 10min after delivery
  identifying the effects of 0.5 µg/kg/h dexmedetomidine for Ramsay sedation scales.(Ramsay standard for evaluation: 1 point: anxious or restless or both; 2 point: cooperative, orientated and tranquil; 3 point: responding to commands; 4 point: brisk response to stimulus; 5 point: sluggish response to stimulus; 6 point: no response to stimulus.)
Placental Transfer of Dexmedetomidine in Epidural | at the delivery of the baby
  identifying the effects of 0.5 µg/kg/h dexmedetomidine for the rate of placental transfer of dexmedetomidine(CUV/CMV).
  Methods:
  When the baby was born, we double clamped the umbilical cord,and extracted 3ml blood from the maternal vein(MV) on the no venous route hand, umbilical artery(UA) and umbilical vein(UV) from the isolated placenta. The blood blood from Dex group were injected heparin sodium anticoagulant tube, centrifuged 3500 revolutions per minute for 5 minutes and separated of plasma to -20℃ frozen preservation. High-performance liquid chromatography-mass spectrometry(HPLC-MS/MS) was then used for measuring the plasma dexmedetomidine concentrations (CUV, CUA and CMV). The rate of placental transfer of dexmedetomidine is CUV/CMV.

CONTACTS AND LOCATIONS:
Overall Officials: Cunming Liu, MD, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes